CLINICAL TRIAL: NCT03757962
Title: Evaluation of Food Additive Contributions to Obesity - Feasibility Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Natalia McInnes, Associate Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5157
Record Dates: First submitted 2018-11-23; First posted 2018-11-29 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Obesity
Keywords: dietary modification
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention (Experimental)
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Limiting dietary exposure to benzoic acid, sorbic acid, polysorbates and related food additives; limiting eating out to a maximum of 2 days per week.

SUMMARY:
The effects of food additives on body weight in humans are largely unknown. This is a before-and-after feasibility study in 5 obese adults who will be followed for 5 months. Eligible participants will meet with the study team and will be taught how to limit the exposure to the studied food additives in their diet. Participants will also be asked to limit eating out to a maximum of 2 days per week. Primary outcomes in this study are recruitment rate, retention rate and adherence to the proposed dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI>/=30 kg/m2
* willingness and ability to follow the proposed dietary intervention
* informed consent

Exclusion Criteria:

* previous or planned bariatric surgery in the next 1 year
* current or planned participation in any structured weight-loss programs in the next 6 months
* current or recent (within the last 6 months) use of weight-loss-inducing drugs or systemic steroids
* bipolar disorder or attention deficit hyperactivity disorder
* current use of anti-depressant or anti-psychotic medications
* eating disorder or any other active disorder that may lead to significant weight changes
* working night shifts
* pregnancy or planned pregnancy in the next 1 year
* uncontrolled diabetes mellitus or diabetes requiring treatment with >2 oral diabetes medications or with insulin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 0 months
Retention rate | 5 months
Adherence to the dietary intervention | 2 to 4 months
  Proportion of meals/beverages suspected to contain the studied food additives on 3 unannounced 24-hour dietary recalls conducted at 2, 3 and 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No